CLINICAL TRIAL: NCT03110601
Title: Trialing of PM Modulation Therapy in Patients With Chronic Intractable Low Back Pain With or Without Leg Pain
Brief Title: Study of PM Modulation Therapy in Trial Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stimgenics LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGEN-2017PM1
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Control - Conventional SCS (Active Comparator): Conventional SCS parameters for 4 days plus/minus 1 day using an external SCS modulator.
  Interventions: Device: Control - Conventional SCS
- Washout Period (No Intervention): 1 day where no stimulation is provided
- Test - Stimgenics SCS (Experimental): Stimgenics SCS parameters for 4 days plus/minus 1 day using an external SCS modulator.
  Interventions: Device: Test - Stimgenics SCS

INTERVENTIONS:
Device: Control - Conventional SCS — Conventional SCS Parameters
  Arms: Control - Conventional SCS
Device: Test - Stimgenics SCS — Stimgenics SCS Parameters
  Arms: Test - Stimgenics SCS

SUMMARY:
Trialing of PM modulation therapy in patients with chronic intractable low back pain

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent to participate in this clinical study based on voluntary agreement after a thorough explanation of the patient's participation is provided to them.
2. Chronic intractable pain of the lower back equal to or greater than pain in lower limbs, and that has been refractory to conservative therapy for ≥ 3 months.
3. Must be older than 18 years old.
4. Average back pain intensity of ≥ 5 out of 10 on the numerical pain rating scale (NPRS).
5. Appropriate candidate for spinal cord stimulation trial.
6. Subjects must be on a stable dose of pain medication regimen for at least 1 month.
7. Female patients who are not pregnant and do not plan to become pregnant during the study. Females of child bearing potential must provide a negative pregnancy test and must be using reliable contraception and must continue to use reliable contraception until study completion. Non-childbearing potential is defined as postmenopausal for at least 2 years or surgical sterilization or hysterectomy at least 3 months before study start. Patients who become pregnant or who have a spouse/significant other that becomes pregnant during the course of this study agree to report pregnancy to the study physician/staff.
8. Must be able to comply with the requirement of study visits and follow-up and phone visits.
9. Have cognitive ability of operate the remote control and follow therapy instructions and directions by clinicians.

Exclusion Criteria:

1. Systemic infection.
2. Any active implanted device.
3. Previous experience with SCS therapy either during a trial or fully implanted
4. Evidence of serious neurological, psychological or psychiatric disorders.
5. Mechanical spinal instability.
6. Patients with uncorrected coagulation disorders or who are on anticoagulation therapy and cannot interrupt the therapy.
7. Patient who are pregnant, breast-feeding or women of childbearing potential with positive pregnancy tests.
8. Human immunodeficiency virus (HIV) infection or a clinically significant infection.
9. Patients who are undergoing or will undergo therapies or diagnostics that involve electromagnetic fields such as: diathermy based therapies, electrocautery, magnetic resonance imaging (MRI), radiofrequency (RF) or microwave ablation, bone growth stimulators, electrolysis, therapeutic ultrasound, ultrasound, lithotripsy, psychotherapeutic procedures, radiation therapy, and transcutaneous electrical nerve stimulation.
10. A clinically significant disorder such as cerebrovascular disease, pulmonary infarction, ischemic heart disease, cardiac dysrhythmia, myocardial infarction, or congestive heart failure or any other as determined by the investigator.
11. Uncontrolled diabetes, uncontrolled pulmonary disease, or uncontrolled hypertension.
12. Patients who have evidence of major psychiatric disease, mental disorder, drug dependency, alcohol dependency, or substance abuse disorders.
13. Patients who have progressive neurological disease such as multiple sclerosis, chronic inflammatory demyelinating polyneuropathy, rapidly progressive arachnoiditis, acute herniated disc, or any other as determined by investigator.
14. Medical condition or pain in other body areas that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study end points.
15. Concurrent participation in another clinical study.
16. Involvement in an injury claim under current litigation or a pending or approved workers' compensation claim.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2017-10-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- StimGenics, Bloomington, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Non-randomized cross-over study in which all eligible participants received the same order of procedures (i.e. Conventional SCS parameters for 4 days, then a washout period of 1 day, then PM-SCS parameters for 4 days).
Groups:
- Single Arm With Multiple Periods: Non-randomized cross-over study in which all eligible participants received the same order of procedures (i.e. Conventional SCS parameters for 4 days, then a washout period of 1 day, then PM-SCS parameters for 4 days).
Period: Conventional SCS Parameters
Arm/Group | Single Arm With Multiple Periods
Started | 25
Completed | 24
Not Completed | 1
Period: Washout Period
Arm/Group | Single Arm With Multiple Periods
Started | 24
Completed | 23
Not Completed | 1
Period: Stimgenics SCS Parameters
Arm/Group | Single Arm With Multiple Periods
Started | 23
Completed | 20
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Chronic Back Pain Patients
Groups:
- Enrolled Patients: Back pain patients that were trialed with Conventional SCS parameters, then after a washout period the same patients were trialed with PM-SCS parameters (Stimgenics SCS parameters).
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Back Pain on Numeric Pain Rating Scale (11-point rating scale) [Mean (Standard Deviation); unit: Score on a scale] — 11-point Numeric Pain Rating Scale (NPRS) with 0 being no pain at all and 10 being the worst pain imaginable (1-3 is rated as mild pain, 4-6 is rated at moderate pain, 7-9 is rated as severe pain). Subject rates average back pain for the past 7 days.
  Score on a scale | 7.4 (1.2)
Leg Pain Numeric Pain Rating Scale (11-point rating scale) [Mean (Standard Deviation); unit: Score on a scale] — 11-point Numeric Pain Rating Scale (NPRS) with 0 being no pain at all and 10 being the worst pain imaginable (1-3 is rated as mild pain, 4-6 is rated at moderate pain, 7-9 is rated as severe pain). Subject rates average leg pain for the past 7 days.
  Score on a scale | 4 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Relative to Baseline and After a Trial Period
Description: Numerical rating pain score measured before and after intervention. 11-point Numeric Pain Rating Scale (NPRS) with 0 being no pain at all and 10 being the worst pain imaginable (1-3 is rated as mild pain, 4-6 is rated at moderate pain, 7-9 is rated as severe pain). Subject rates average pain for the past 7 days.
Time Frame: Baseline and 4 days plus or minus 1 days
Population: Chronic Back Pain Patients with or without leg pain; 4 subjects experience known adverse events (such as lead migration) that prevented them from testing Stimgenics SCS.
Measure: Mean (Standard Deviation); unit: Score on a 11 point scale
Groups:
- Conventional SCS: Mean Back Pain Score after treatment Conventional SCS parameters
- Stimgenics SCS: Mean Back Pain Score after treatments with Stimgenics SCS parameters
Arm/Group | Conventional SCS | Stimgenics SCS
Number analyzed (Participants) | 24 | 20
Score on a 11 point scale | 4.2 (2.0) | 2.4 (1.8)

ADVERSE EVENTS:
Time Frame: 1-10 days
Description: Same as clinicaltrials.gov definition
Groups:
- Conventional SCS: Conventional SCS parameters for 4 days
- Washout Period: Washout period of 1 day
- Stimgenics SCS: Stimgenics SCS parameters for 4 days
Arm/Group | Conventional SCS | Washout Period | Stimgenics SCS
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 3/25 | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional SCS (N=25) | Washout Period (N=20) | Stimgenics SCS (N=20)
Epidural abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional SCS (N=25) | Washout Period (N=20) | Stimgenics SCS (N=20)
Lead movement (Surgical and medical procedures) | 3 (3) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Patients were evaluated during the trial phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT03110601/Prot_SAP_000.pdf